CLINICAL TRIAL: NCT00837447
Title: Range of Motion of Standard and High-Flexion Posterior Cruciate Retaining Total Knee Prostheses A Prospective, Randomized Study
Brief Title: Range of Motion of Standard and High-Flexion Posterior Cruciate Retaining Total Knee Prostheses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor and Director, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-7
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NexGen CR knee prosthesis (Active Comparator): side of knee operated with total knee replacement with Nexgen CR prosthesis
  Interventions: Device: Total knee replacement with NexGen CR knee prosthesis
- NexGen CR-Flex knee prosthesis (Active Comparator): side of knee operated with total knee arthroplasty using Nexgen CR-flex prosthesis
  Interventions: Device: Total knee replacement(TKR) with Nexgen CR-flex

INTERVENTIONS:
Device: Total knee replacement with NexGen CR knee prosthesis — comparison of functional outcome in patients receiving either NexGen posterior cruciate-retaining or a high-flexion posterior cruciate-retaining total knee prosthesis
  Other Names: NexGen CR
  Arms: NexGen CR knee prosthesis
Device: Total knee replacement(TKR) with Nexgen CR-flex — TKR using Nexgen CR-flex implant
  Other Names: Nexgen CR-flex
  Arms: NexGen CR-Flex knee prosthesis

SUMMARY:
The purpose of this prospective, randomized study was to compare pain, functional outcome and ranges of motion of the knees in patients receiving either a standard posterior cruciate-retaining or a high-flexion posterior cruciate-retaining total knee prosthesis.

DETAILED DESCRIPTION:
The main goals of total knee arthroplasty are pain relief and improvement of function and range of motion. The purpose of this study was to compare ranges of motion of the knees in patients receiving either a standard posterior crucaite-retaining or a high-flexion posterior cruciate-retaining total knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis that was severe enough to warrant total knee arthroplasty after an adequate trial of nonoperative therapy, and the need for bilateral total knee arthroplasties

Exclusion Criteria:

* inflammatory arthritis
* osteoarthritis of the hip causing pain or restricted mobility
* a foot or ankle disorder which limited walking
* dementia or a neurological disorder including a past history of stroke which affected mobility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University Mokdong Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- NexGen CR and CR-flex Knee Prosthesis: The NexGen posterior cruciate-retaining total knee arthroplasty prosthesis (NexGen CR Prosthesis; Zimmer)) on one side and The NexGen posterior cruciate-retaining flex total knee arthroplasty prosthesis (NexGen CR-Flex; Zimmer) on the other side
Period: Overall Study
Arm/Group | NexGen CR and CR-flex Knee Prosthesis
Started | 54 (Each of the 54 pts received a Nexgen CR on one side and a Nexgen CR-Flex on the contralateral side.)
Completed | 54 (Each of the 54 pts received a Nexgen CR on one side and a Nexgen CR-Flex on the contralateral side.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NexGen CR and CR-flex Knee Prosthesis
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 5
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Society Knee Score
Description: change in knee score will be compared with baseline and follow up of 3 years. The knee society knee score range from 0 to 100 points, 100 being the best possible outcome.
  Baseline-NexGen (CR) knee socre:29 points Baseline-NexGen (CR-Flex) knee socre:29 points Follow up of 3 years-NexGen (CR) knee socre: 93.7 points Follow up of 3 years-NexGen (CR-Flex) knee socre: 93.9 points
Time Frame: baseline and 3 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Flexion Posterior Cruciate Retaining TKA | High-Flexion Posterior Cruciate Scrificing TKA
Number analyzed (Participants) | 54 | 54
scores on a scale | 93.9 (4.66) | 93.7 (4.53)

ADVERSE EVENTS:
Arm/Group | NexGen CR and CR-flex Knee Prosthesis
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

LIMITATIONS AND CAVEATS:
First, the knee scoring system is prone to intraobserver variability. Second, we had no interobserver variability and this could have lead to bias in interpreting radiographic results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No